CLINICAL TRIAL: NCT04979975
Title: A Randomized, Single-blind, Placebo-control, Parallel, Phase II Trial to Evaluate the Safety and Efficacy of UB-621 in Adults With Recurrent Genital HSV-2 Infection
Brief Title: Evaluating Safety and Efficacy of Repeat Doses of UB-621in Adult Patients With Recurrent Genital Herpes
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UBP Greater China (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBP-A229-HSV
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Recurrent Genital Herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Experimental): placebo matching UB-621
  Interventions: Other: Placebo
- UB-621 low-dose (Experimental): low-dose of UB-621
  Interventions: Biological: UB-621 low-dose
- UB-621 high-dose (Experimental): high-dose of UB-621
  Interventions: Biological: UB-621 high-dose

INTERVENTIONS:
Other: Placebo — PBO- placebo matching to UB-621
  Arms: Placebo
Biological: UB-621 low-dose — fully human anti-HSV mAb
  Arms: UB-621 low-dose
Biological: UB-621 high-dose — fully human anti-HSV mAb
  Arms: UB-621 high-dose

SUMMARY:
To evaluate the efficacy of repeat-dose UB-621 for the recurrent genital HSV-2 infection To evaluate the safety and tolerance of repeat-dose UB-621 for the recurrent HSV-2 infection To evaluate the pharmacokinetics of repeat-dose UB-621 in RGH patients

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧18 years at the time of signing ICF
2. HSV-2 seropositive when screening
3. A history of recurrent genital herpes and experience 6-12 episodes in the past year
4. Negative result of the HIV assay
5. In baseline period, subject have to present at the site within 72 hours after the occurrence of new lesions
6. Keep daily diary during the study period
7. Female subjects: negative serum β-HCG at screening and no beast-feeding.
8. Use contraception during study participation
9. Understanding and willing to fully comply with study interventions and restrictions.

Exclusion Criteria:

1. Any medical conditions that may interfere the assessment of UB-621efficacy, or any medical conditions that may present symptoms in the anogenital regions (such as syphilis, genital warts).
2. History of malignancy, diabetes, auto-immune diseases or immunodificiency diseases.
3. Use of systemic steroids or immunomodulators within 30 days prior to the screening
4. Participating any clinical trials within 30 days prior to the screening, or within 5 half-life of any investigational drugs, take the longer.
5. Vaccination within 30 days prior to the screening.
6. Prior exposure to any HSV vaccines
7. Known hypersensitive to monoclonal antibodies
8. ECG abnormalities with clinical relevance or cardiovascular diseases at screening
9. Serum creatinine > 1.5 mg/dL at screening
10. AST and ALT > 2.5 x ULN at screening
11. HBsAg positive or HCT antibody positive at screening
12. Syphilis RPR test positive at screening
13. TB history or documented T-spot positive, or now is under treatment of TB
14. Any other circumstances that are determined to affect the conduct or successful completion of the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to first recurrence | 26 weeks
  Time to first recurrence episode after experimental drug administration as reported by patient and verified by investigator.

SECONDARY OUTCOMES:
Proportion of subjects with episodes | 26 weeks
  Proportion of subjects with episodes is calculated as the number of subjects with episodes divided by the number of total subjects.
Lesion rate | 26 weeks
  Lesion rate is calculated as the number of days with lesion divided by the number of study days.
Duration of recurrent lesions | 26 weeks
  Duration of recurrent lesions is calculated as consecutive days with lesions.
Recurrence rate | 26 weeks
  Recurrence rate is defined as number of recurrences divided by the total number of study days.

OTHER OUTCOMES:
HSV-2 shedding rate | 12 weeks
  Viral shedding rate is defined as the number of positive anogenital swabs divided by total number of swabs.
Clinical and Subclinical HSV-2 Shedding Rates | 12 weeks
  Daily record of subject self-assessment of genital lesions in subject diary in addition to anogenital swabs collected daily from subjects during the follow-up periods will be used to evaluate the clinical (lesional) and subclinical (non-lesional) HSV-2 shedding rates.
Rate of HSV-2 Shedding Episodes | 12 weeks
  The rate of HSV-2 shedding episodes is the number of onsets of shedding episodes divided by the total number of days with swabs collected. Shedding episodes are defined as consecutive HSV-2 positive swab results including no more than 1 consecutive negative result or missed swab. The episodes are preceded and followed by 2 consecutive negative swab results.
HSV-2 viral load | 12 weeks
  Anogenital swab samples collected from subjects during follow-up period will be used to quantify HSV-2 DNA copies.